CLINICAL TRIAL: NCT06512766
Title: Cicatricial Alopecia: a Retrospective Study on the Systemic Treatment of Lichen Planopilaris and Frontal Fibrosing Alopecia
Brief Title: a Retrospective Study on the Systemic Treatment of LPP and FFA
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, DirkJan Hijnen, MD, PhD, Erasmus Medical Center
Other Study IDs: 9434
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cicatricial Alopecia; Lichen Planopilaris; Lichen Plano-Pilaris; Frontal Fibrosing Alopecia; Hair Diseases; Scarring Alopecia; Hair Loss/Baldness
Keywords: Systemic treatment
MeSH Terms: conditions — Alopecia; Lichen Planus; Hair Diseases | interventions — Hydroxychloroquine; Methotrexate; Cyclosporine; Retinoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lichen planopilaris: Patients in this group were diagnosed and treated for lichen planopilaris (LPP), a form of primary lymphocytic cicatricial alopecia. Treatment options included hydroxychloroquine (HCQ), methotrexate (MTX), cyclosporine A (CsA), and retinoids. The effectiveness of these treatments varied among patients. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments were not consistent.
  Interventions: Drug: Hydroxychloroquine; Drug: Methotrexate; Drug: Cyclosporine A; Drug: Retinoids
- Frontal fibrosing alopecia: Patients in this group were diagnosed and treated for frontal fibrosing alopecia (FFA), a form of primary lymphocytic cicatricial alopecia. Treatment options included hydroxychloroquine (HCQ), methotrexate (MTX), cyclosporine A (CsA), and retinoids. The effectiveness of these treatments varied among patients. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments were not consistent.
  Interventions: Drug: Hydroxychloroquine; Drug: Methotrexate; Drug: Cyclosporine A; Drug: Retinoids

INTERVENTIONS:
Drug: Hydroxychloroquine — Patients in this group were treated with hydroxychloroquine (HCQ), a systemic medication commonly used as a first-line treatment due to its ease of use and established safety profile. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments varied among patients.
Drug: Methotrexate — This group consists of patients treated with methotrexate (MTX), a systemic medication often used as a second-line treatment for its effectiveness in reducing inflammation and controlling autoimmune responses. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments varied among patients.
Drug: Cyclosporine A — Patients in this group were treated with cyclosporine A (CsA), a potent immunosuppressive agent used for its effectiveness in controlling severe inflammatory responses. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments varied among patients.
Drug: Retinoids — This cohort includes patients treated with retinoids, which are used for their ability to modulate cell growth and differentiation. Due to the retrospective nature of the study, the dosage form, dosage, frequency, and duration of treatments varied among patients.

SUMMARY:
This retrospective study aims to assess the effectiveness of systemic treatments for lichen planopilaris (LPP) and frontal fibrosing alopecia (FFA) in patients treated at the Erasmus MC University Medical Center. LPP and FFA are chronic inflammatory hair disorders leading to irreversible hair loss. The study evaluates treatment responses to systemic medications, including hydroxychloroquine, methotrexate, cyclosporine A, and retinoids.

DETAILED DESCRIPTION:
Cicatricial alopecia, also known as scarring alopecia, refers to a group of rare chronic inflammatory hair disorders resulting in irreversible hair loss. Lichen planopilaris (LPP) and frontal fibrosing alopecia (FFA) are the most common forms of primary lymphocytic cicatricial alopecia, affecting predominantly postmenopausal women. These conditions lead to significant quality of life impairment due to their chronic nature and the lack of effective, standardized treatment protocols. The study aimed to address the gap in evidence-based treatment guidelines by investigating the effectiveness of various systemic therapies currently used in clinical practice. The retrospective cohort study reviewed medical records of patients diagnosed with LPP or FFA at the Department of Dermatology, Erasmus MC University Medical Center, from July 2016 to July 2022.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LPP or FFA
* 18 years or older

Exclusion Criteria:

* Other forms of cicatricial alopecia than LPP or FFA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with International Classification of Diseases and Related Health Problems, Tenth Revision (ICD-10) diagnosis: L66 cicatricial alopecia, between July 2016 and July 2022, from the Department of Dermatology, Erasmus MC University Medical Center, were included.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Treatment response | The time frame for evaluating treatment response varies per patient due to the retrospective nature of the study. Patients were treated and assessed at various intervals between July 2016 and July 2022.
  The primary outcome measure is the treatment response of systemic treatment options in patients diagnosed with LPP and FFA. Treatment response is categorized into three groups: no response (progression of symptoms, hair loss, and trichoscopic activity), moderate response (improvement in symptoms, reduced hair loss progression, or reduction in trichoscopic activity), and good response (absence of symptoms, no further hair loss, and no trichoscopic activity).

SECONDARY OUTCOMES:
Reason for discontinuation | The time frame for evaluating reason for discontinuation varies per patient due to the retrospective nature of the study. Patients were treated and assessed at various intervals between July 2016 and July 2022.
  This secondary outcome measure assesses the discontinuation rates of systemic treatments (HCQ, MTX, CsA, and retinoids) and the reasons for discontinuation, such as side effects or insufficient treatment effects.

CONTACTS AND LOCATIONS:
Overall Officials: DirkJan Hijnen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided